CLINICAL TRIAL: NCT04175080
Title: Clinical Significance and Diagnosis of Sarcopenia in Patients With Heart Failure With Preserved Ejection Fraction
Brief Title: Clinical Significance and Diagnosis of Sarcopenia in Cardiac Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Agata Bielecka-Dabrowa, MD, PhD, Department of Hypertension, Principal Investigator, Medical University of Lodz
Other Study IDs: RNN/80/17/KE
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Hypertension; Sarcopenic Obesity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control
- HFpEF group
- Hypertensive group: Patients in which the results of BNP/NT-proBNP did not confirm the diagnosis of HFpEF were classified as hypertensive group.

SUMMARY:
Obesity sarcopenia, characterized by the coexistence of excess fat and muscle mass reduction, may contribute to the pathophysiology of exercise intolerance in patients with heart failure with preserved ejection fraction (HFpEF). The project will examine the impact of selected circulating miRNAs on processes that may form the pathophysiological basis for HFpEF development and obesity sarcopenia in correlation with biochemical markers, echocardiographic assessment and non-invasive assessment of hemodynamic parameters. In addition, the impact of LDL and HDL on these diseases will be assessed. Determinations of selected adipokines and asymmetric dimethylarginine will also be carried out and their effects on the cardiovascular system will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* control group: healthy volunteers
* study groups: patients with HFpEF. Patients in which the results of BNP/NT-proBNP did not confirm the diagnosis of HFpEF were classified as hypertensive group.

Exclusion Criteria:

* coronary artery disease
* unstable hypertension
* heart failure class IV NYHA
* condition after percutaneous or surgical revascularization
* pulmonary hypertension in echocardiography
* obstructive or restrictive lung diseases
* congenital heart disease
* arrhythmias (including atrial fibrillation)
* pacemaker or implantable cardioverter defibrillator
* hyperthyroidism or hypothyroidism
* pregnancy or lactation
* hemodynamically significant acquired heart defects
* cardiomyopathies
* GFR <60 ml/min/1.73 m2
* other medical conditions such as: cancer, significant anemia, diabetes, alcohol and drug abuse, chronic inflammatory diseases and other
* the patient's inability to cooperate and / or give informed consent to participate in the study

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults in the age 35-70. Patients will be recruited from the patients of Cardiology Outpatient Clinic and Nephrology, Hypertension and Family Medicine Clinic of the University Clinical Hospital WAM - Central Veterans Hospital in Łódź
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
The level of biochemical parameters | through study completion, an average of 1 year
Left ventricular systolic and diastolic function | through study completion, an average of 1 year
Arterial stiffness | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Agata Bielecka-Dąbrowa, MD, PhD, Principal Investigator — Department of Hypertension Medical University of Lodz
Locations (1):
- Department of Hypertension MU of Lodz, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paduszynska A, Sakowicz A, Banach M, Maciejewski M, Dabrowa M, Bielecka-Dabrowa A. Cardioprotective properties of leptin in patients with excessive body mass. Ir J Med Sci. 2020 Nov;189(4):1259-1265. doi: 10.1007/s11845-020-02211-9. Epub 2020 Mar 20. PMID 32198598